CLINICAL TRIAL: NCT01310959
Title: Establishing a Data Base for Aplastic Anemia and Other Marrow Failure Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2021-084; RAC# 2021-084
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Aplastic Anemia and Other Marrow Failure Syndrome
Keywords: Aplastic Anemia Marrow Failure Syndrome
MeSH Terms: conditions — Anemia, Aplastic | interventions — Database Management Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Database — Database

SUMMARY:
Establishing a Data Base for Aplastic Anemia and Other Marrow Failure Syndrome

DETAILED DESCRIPTION:
Establishing a Data Base for Aplastic Anemia and Other Marrow Failure Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed Aplastic Anemia and Other Marrow Failure Syndrome Database.

Exclusion Criteria:

* Patients with diagnosis other than Aplastic Anemia and Other Marrow Failure Syndrome Database.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Aplastic Anemia and Other Marrow Failure Syndrome Database
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: H Al-Zahrani, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia